CLINICAL TRIAL: NCT06175611
Title: Clinical Performance Study for EDAN's COVID-19/Flu A/Flu B/RSV Test Kits on Subjects Suspected of Respiratory Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: EDAN Instruments Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL30_2023_08
Record Dates: First submitted 2023-12-18; First posted 2023-12-19 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: SARS-CoV2 Infection; Influenza A; Influenza B; Respiratory Syncytial Virus (RSV)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Anterior nasal and oropharyngeal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Site 1. Laboratorio Central Health Diagnostics Quirónsalud: COVID-19/Flu A/Flu B/RSV Test Kit
  Interventions: Device: COVID-19/Flu A/Flu B/RSV Test Kit
- SIte 2. Hospital General Universitario Dr. Balmis de Alicante: COVID-19/Flu A/Flu B/RSV Test Kit
  Interventions: Device: COVID-19/Flu A/Flu B/RSV Test Kit
- Site 3. Hospital Universitario de Getafe: COVID-19/Flu A/Flu B/RSV Test Kit
  Interventions: Device: COVID-19/Flu A/Flu B/RSV Test Kit

INTERVENTIONS:
Device: COVID-19/Flu A/Flu B/RSV Test Kit — The performance characteristics of EDAN's Test Kit will be evaluated in a prospective, non-randomized, observational, post-market, multicenter, comparison clinical performance study using anterior nasal and oropharyngeal swabs from subjects suspected of respiratory infection.
  Samples will be obtained fresh, collected prospectively and will be tested with the study device COVID- 19/Flu A/Flu B/RSV Test Kit. The results will be compared against a reference, CE marked, in-vitro diagnostic device, used in the standard of care.
  This clinical performance study has been designed to minimize any possible, discomfort, or other foreseeable risks to the participants.

SUMMARY:
The primary objective of this clinical performance study is to evaluate and further validate the clinical performance of:

1. ClariLight Influenza A/B & SARS-CoV-2 test kits and
2. ClariLight Influenza A/B & RSV test kits, for the qualitative detection and differential diagnosis of SARS-CoV-2, influenza A, influenza B, and respiratory syncytial virus (RSV) present in anterior nasal and oropharyngeal swab, in combination with an automated molecular diagnostic analyzer and sample collection tube by comparing them against a CE marked, in-vitro diagnostic device, used in the standard of care.

DETAILED DESCRIPTION:
Prospective, non-randomized, observational, post-market, multicenter, clinical performance study using anterior nasal and oropharyngeal swabs from subjects suspected of respiratory infection for evaluating the clinical performance of ClariLight Influenza A/B & SARS-CoV-2 Cartridge and the ClariLight Influenza A/B & RSV Cartridge by comparing them against a reference standard of care, CE marked, comparator device.

This clinical performance study has been designed to minimize any possible, discomfort, or other foreseeable risks to the participants.

This clinical performance study:

1. Does not involve surgically invasive sample-taking
2. Is not interventional as test results will not influence patient management decisions neither they will be used to guide treatment
3. There are no additional invasive procedures or other risks for the subjects. The device is being used within the scope of its CE marked intended purpose and for the specimen types claimed which include standard of care specimen collection procedures.

No specific follow-up of subjects providing swabs is required following termination, temporary suspension or early termination of the study, or withdrawal of the subject's informed consent. The participation of each subject for the total duration of the study will amount to 1 hour, finishing the participation in day 1. Subjects will be provided with the Investigator's contact information and be instructed to contact the Investigator if they experience any complications from the specimen collection procedures within twenty-four (24) hours of the visit".

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL the inclusion criteria described below to be eligible for this clinical performance study.

1. Subjects with suspected respiratory infection who have physical signs/symptoms, such as chills, fever, headache, myalgia, fatigue, nasal congestion, sore throat, and other symptoms.
2. Subjects able to provide anterior nasal swabs and oropharyngeal swabs for testing on the study device according to the instructions for use of that device.
3. Subjects able to provide comparator samples according to the instructions for use of the comparator device.
4. Subjects able to provide study and comparator samples within 24 hours to allow for a valid comparison.
5. Subjects or their legal guardians willing and able to provide written informed consent.

Exclusion Criteria:

Subjects who meet any of the exclusion criteria described below will NOT be eligible for this clinical performance study.

1. Subjects who have undergone anterior nasal, or oropharyngeal sampling within the past 30 minutes (i.e. a minimum wait of 30 minutes is required before collecting swabs for the study device if previous anterior nasal or oropharyngeal samples were collected from the same subject).
2. Subjects or their legal guardians unwilling and unable to provide informed consent.
3. Subjects who have had a nasal wash or aspirate procedure within the past 24 hours.
4. Women who are pregnant or currently breastfeeding.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises of subjects suspected of respiratory infection by their healthcare provider who meet the all the inclusion criteria and none of the exclusion criteria detailed in the CPSP.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Positive Percentage Agreement (PPA) | Day 1. No follow-up is required for this study.
  The PPA is defined as the proportion of positive results from the comparator or reference method that are correctly identified as positive by study device. PPA will be determined across all swab types tested (anterior nasal swab and oropharyngeal) against the standard of care comparator (NAAT and sequencing where appropriate) for all targets individually. Values will be estimated, with corresponding 2-sided 95% score confidence intervals (CIs).
Negative Percentage Agreement (NPA). | Day 1. No follow-up is required for this study.
  The NPA is defined as the as the proportion of negative results from the comparator or reference method that are correctly identified as negative by the study device.
  NPA will be determined across all swab types tested (anterior nasal swab and oropharyngeal) against the standard of care comparator (NAAT and sequencing where appropriate) for all targets individually. Values will be estimated, with corresponding 2-sided 95% score confidence intervals (CIs).

SECONDARY OUTCOMES:
Rate of adverse events, serious adverse events and device deficiencies leading to a serious adverse event. | Day 1. No follow-up is required for this study. Nevertheless, subjects who have undergone sample collection can contact the study's Principal Investigator throughout the whole clinical performance study.
  Rate of adverse events that occur during the clinical performance study and that are critical to the evaluation of the study results.
  Rate of serious adverse events that have a causal relationship with the device, the comparator, or the study procedure or where such causal relationship is reasonably possible.
  Rate of device deficiencies that occur during the clinical performance study, which might have led to a serious adverse event, if appropriate action had not been taken, intervention had not occurred, or circumstances had been less fortunate.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital General Universitario Dr. Balmis de Alicante, Alicante
  - Laboratorio Central Health Diagnostics Quirónsalud, Madrid
  - Hospital Universitario de Getafe, Madrid

IPD SHARING:
Plan to Share IPD: No